CLINICAL TRIAL: NCT04750525
Title: A Non-invasive Intervention (BreEStim) for Management of Phantom Limb Pain (PLP) After Limb Amputation
Brief Title: A Non-invasive Intervention (BreEStim) for Management of Phantom Limb Pain (PLP) After Limb Amputation (Experiment 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sheng Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-20-1032 (Experiment 1)
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Pain Management
Keywords: Phantom Limb Pain; BreEStim
MeSH Terms: conditions — Agnosia; Phantom Limb

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BreEStim 120, then EStim 120 (Experimental): BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation. EStim is transcutaneous electrical nerve stimulation.
  Interventions: Device: BreEStim; Device: EStim
- EStim 120, then BreEStim 120 (Experimental): BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation. EStim is transcutaneous electrical nerve stimulation.
  Interventions: Device: BreEStim; Device: EStim

INTERVENTIONS:
Device: BreEStim — 120 BreEStim stimuli will applied for about 10-30 minutes.
Device: EStim — 120 EStim stimuli will applied for about 10-30 minutes.

SUMMARY:
The purpose of this study is to compare the effectiveness of innovative intervention of breathing controlled electrical stimulation (BreEStim) and conventional electrical stimulation (EStim) in management of neuropathic phantom limb pain in patients after limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* has phantom limb pain (PLP) after amputation of one limb, upper or lower limb;
* has chronic pain, >3 months;
* is stable on oral pain medications at least two weeks. (patients are allowed to continue their pain medications, i.e., no change in pain medications.)

Exclusion Criteria:

* currently adjusting oral pain medications for their PLP;
* has pain, but not PLP (e.g., from inflammation at the incision wound of the residual limb);
* has a pacemaker, or other metal and/or implanted devices;
* has cognitive impairment from brain injury or are not able to follow commands, or to give consent;
* has amputation in multiple limbs;
* have asthma or other pulmonary diseases;
* are not medically stable;
* have preexisting psychiatric disorders;
* alcohol or drug abuse;
* have a history of seizures/Epilepsy, or taking benzodiazepines, anticonvulsants, and antidepressants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (15-30 Minutes)
Arm/Group | BreEStim 120, Then EStim 120 | EStim 120, Then BreEStim 120
Started | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0
Period: Washout (About 3-14 Days)
Arm/Group | BreEStim 120, Then EStim 120 | EStim 120, Then BreEStim 120
Started | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0
Period: Second Intervention (15-30 Minutes)
Arm/Group | BreEStim 120, Then EStim 120 | EStim 120, Then BreEStim 120
Started | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 participants were assigned to the EStim 120, then BreEStim 120 arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | BreEStim 120, Then EStim 120 | EStim 120, Then BreEStim 120 | Total
Number analyzed (Participants) | 15 | 0 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 13 |  | 13
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  | 5
  Male | 10 |  | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 6 |  | 6
  Black or African American | 6 |  | 6
  Hispanic or Latino | 2 |  | 2
  Asian | 0 |  | 0
  Others | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level as Measured by the Visual Analog Scale (VAS).
Description: VAS scores are recorded from 0 to 10 with 0 being "no pain" and 10 being "worst pain", a higher score indicating a higher level of pain. Change is reported as [(VAS score at baseline) - (VAS Score 10 minutes after intervention)] - a positive value indicates that the score (and pain level) decreased
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BreEStim 120: BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation. 120 BreEStim stimuli will applied for about 10-30 minutes.
- EStim 120: EStim is transcutaneous electrical nerve stimulation. 120 EStim stimuli will applied for about 10-30 minutes.
Arm/Group | BreEStim 120 | EStim 120
Number analyzed (Participants) | 15 | 15
score on a scale | 1.38 (1.24) | 1.27 (1.13)

2. Secondary Outcome: Change in Sensation Threshold on Amputated Limb Measured by Electrical Sensation Threshold (EST)
Description: Electrical Sensation Threshold (EST) is the minimum electrical current intensity that a person can reliably perceive as a sensation on their skin. This threshold is self-reported by the subjects, and electrical intensity values are recorded when participants first detect the electrical stimulation. Change is reported as [(EST at 5 minutes after intervention) - (EST at baseline)] - a positive value indicates a decrease in sensation perception.
Time Frame: Baseline, 5 minutes after intervention
Measure: Mean (Standard Deviation); unit: milliampere (mA)
Groups:
- BreEStim 120 Treatment: BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation. 120 BreEStim stimuli will applied for about 10-30 minutes
- EStim 120 Treatment: EStim is transcutaneous electrical nerve stimulation. 120 EStim stimuli will applied for about 10-30 minutes.
Arm/Group | BreEStim 120 Treatment | EStim 120 Treatment
Number analyzed (Participants) | 15 | 15
milliampere (mA) | 1.00 (4.34) | 0.44 (2.58)

3. Secondary Outcome: Change in Pain Threshold on Amputated Limb Measured by Electrical Pain Threshold (EPT)
Description: An Electrical Pain Threshold (EPT) refers to the minimum intensity of electrical stimulation required to produce a perceptible pain sensation on a person's skin, essentially measuring the point at which an electrical current becomes painful. The EPT is self-reported by subjects when they feel the electrical intensity begins to cause pain. Change is reported as [(EPT at 5 minutes after intervention) - (EPT at baseline)] - a positive value indicates an increase in pain threshold.
Time Frame: Baseline, 5 minutes after intervention
Measure: Mean (Standard Deviation); unit: milliampere (mA)
Arm/Group | BreEStim 120 Treatment | EStim 120 Treatment
Number analyzed (Participants) | 15 | 15
milliampere (mA) | 3.99 (19.18) | 3.39 (7.14)

4. Other Pre Specified Outcome: Difference in Heart Rate Variability (HRV) Measured by Electrocardiogram (ECG)
Description: HRV is a measure of the variation in time between each heartbeat. We use HRV to identify the autonomic nervous system changes after intervention treatment. A 5-minute HRV will be recorded prior to the intervention, and 10 mins after the intervention. In this study, the major HRV outcome measurement parameters we choose include: SDNN (standard deviation of normal-to-normal intervals), RMSSD (root mean square of successive differences), and pNN50 (percentage of adjacent RR intervals differing by more than 50ms). SDNN represents the overall variability in the time intervals between heartbeats, providing a general measure of autonomic nervous system function. RMSSD primarily reflects short-term variations in heart rate, often considered a good indicator of parasympathetic activity. pNN50 Measures the proportion of consecutive heartbeats with a significant difference in interval, reflecting the instantaneous changes in heart rate and parasympathetic activity and modulation.
Time Frame: Baseline, 10 minutes after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | BreEStim 120 | EStim 120
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BreEStim 120 (N=15) | EStim 120 (N=15)
Redness (Skin and subcutaneous tissue disorders) | 4 | 4
discomfort (General disorders) | 15 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT04750525/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT04750525/ICF_001.pdf